CLINICAL TRIAL: NCT06012708
Title: An Open-label, Dose-escalation and Dose-finding, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of KN510, KN713 as Combination Therapy in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of KN510, KN713
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Cancer Cure-Bio Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCCKN-101
Record Dates: First submitted 2023-08-04; First posted 2023-08-25 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Experimental)
  Interventions: Drug: KN510 60mg/day + KN713 60mg/day
- Dose Level 2 (Experimental)
  Interventions: Drug: KN510 120mg/day + KN713 60mg/day
- Dose Level 3 (Experimental)
  Interventions: Drug: KN510 120mg/day + KN713 90mg/day
- Dose Level 4 (Experimental)
  Interventions: Drug: KN510 120mg/day + KN713 120mg/day

INTERVENTIONS:
Drug: KN510 60mg/day + KN713 60mg/day — Once daily with 28 days (4 weeks) as one cycle.
  Arms: Dose Level 1
Drug: KN510 120mg/day + KN713 60mg/day — Once daily with 28 days (4 weeks) as one cycle.
  Arms: Dose Level 2
Drug: KN510 120mg/day + KN713 90mg/day — Once daily with 28 days (4 weeks) as one cycle.
  Arms: Dose Level 3
Drug: KN510 120mg/day + KN713 120mg/day — Once daily with 28 days (4 weeks) as one cycle.
  Arms: Dose Level 4

SUMMARY:
To evaluate the safety and tolerability of the combination therapy of KN510 and KN713 and determine the MTD and RP2D in patients with advanced solid tumors.

DETAILED DESCRIPTION:
It is expected that KN510 and KN713 will broaden the range of target patient groups and overcome resistance to the drugs in an innovative manner by targeting the common metabolic process of cancer cells, unlike existing targeted therapies whose application is limited depending on the presence of specific mutation and combination of mutations as they mainly target a single tyrosine kinase.

In this study, the safety and tolerability of combination therapy of KN510 and KN713, including the dose limiting toxicity (DLT) and maximum tolerated dose (MTD), will be evaluated in patients with advance solid tumors and based on this, the recommended phase 2 dose (RP2D) will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 19-75 years
2. Unresectable advanced or metastatic solid tumors that are confirmed as progressive disease (PD) after the standard of care currently known to have clinical benefits, or for which no currently available standard therapies exist due to intolerance, ineligibility, rejection, etc.
3. At least one measurable lesion per RECIST ver1.1
4. The Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
5. Life expectancy of at least 12 weeks
6. Confirmed adequate hematologic, renal, and hepatic functions according to the following criteria (Laboratory tests may be repeated once during the screening period):

   A. Hematological function
   * Absolute neutrophil count (ANC) ≥1,500/μL
   * Hemoglobin ≥9 g/dL
   * Platelet count ≥100,000/μL

   B. Renal function: Creatinine clearance (CrCl*) >60 mL/min

   *Cockcroft-Gault equation

   C. Hepatic function
   * Aspartate aminotransferase (AST) ≤3.0 × ULN
   * Alanine aminotransferase (ALT) ≤3.0 × ULN (AST/ALT ≤5 × ULN, if hepatic metastasis is confirmed)
   * Total bilirubin ≤1.5 × ULN (with the exception of confirmed Gilbert's syndrome)

   D. Coagulation function: Prothrombin time international normalized ratio (PT INR) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN
7. Voluntary written consent to participate in this study

Exclusion Criteria:

1. Hypersensitivity to the active ingredient or excipients of KN510 or KN713
2. Any of the following medical (surgical) history or comorbidities at the screening visit:

   A. Major surgery that requires general anesthesia or a respiratory assist device within 4 weeks prior to screening (within 2 weeks for video-assisted thoracoscopic surgery [VATS] or open-and-closed [ONC] surgery)

   B. Clinically significant arrhythmia, acute myocardial infarction, unstable angina, or NYHA Grade Ⅲ or Ⅳ heart failure within 24 weeks prior to screening

   C. Pulmonary thrombosis, deep vein thrombosis, or bronchial asthma, obstructive pulmonary disease or other life-threatening severe lung disorder (e.g., acute respiratory distress syndrome, lung failure) considered ineligible for participation in the study within 24 weeks prior to screening

   D. Grade 3 or higher active infectious conditions which require systemic antibiotics, antivirals, etc. within 2 weeks prior to screening

   E. Clinically significantly symptomatic or uncontrolled central nervous system or brain metastases at screening (except for patients who have discontinued systemic corticosteroid treatment at least 4 weeks prior to baseline and have been stable for at least 4 weeks)

   F. Hematologic malignancy including lymphoma at screening

   G. Uncontrolled hypertension (systolic blood pressure [SBP]/diastolic blood pressure [DBP] ≥160/100 mmHg) at screening

   H. Parkinson's disease, parkinsonian symptoms, tremors, restless leg syndrome, and other related movement disorders at screening

   I. Active hepatitis B* or C† at screening

   * Defined as HBsAg positive at screening; patients on stable antiviral regimen may participate

   † Defined as HCV Ab positive at screening; patients who test negative for HCV RNA may participate

   J. Known human immunodeficiency virus (HIV) infection

   K. Difficulty (e.g., problem swallowing) in oral administration of KN510 and KN713 or disease (celiac disease, Crohn's disease, or intestinal resection which is clinically significant or impacts absorption) which impacts absorption at screening

   L. History or suspected symptoms of gastroesophageal reflux disease (GERD) such as gastric ulcer, duodenal ulcer, and reflux esophagitis at screening

   M. History of autoimmune diseases at screening

   N. Deemed ineligible for the study for having a comorbidity that is uncontrolled or requires treatment
3. Prior treatment with any of the following medications within 2 weeks prior to screening

   A. Proton pump inhibitors (PPIs) other than the IP

   B. Strong CYP2C19 inducers: Rifampicin, Apalutamide, Rifamycin, Rifaximin, Rifapentine

   C. Strong CYP2C19 inhibitors: Fluvoxamine, Ticlopidine, Chloramphenicol, Delavirdine, Gemfibrozil, Stiripentol, Fluoxetine, Imipramine, Clomipramine, Lansoprazole, Isoniazid, Zafirlukast, Tioconazole, Miconazole

   D. CYP2C19 substrates: Clopidogrel, Citalopram, Cilostazol, Phenytoin, Diazepam

   E. Vitamin K antagonists: Warfarin, Dicoumarol, Phenindione, Phenprocoumon, Acenocoumarol, Ethyl biscoumacetate, Fluindione, Clorindione, Diphenadione, Tioclomarol

   F. Antiretrovirals: Rilpivirine-containing products, Atazanavir, Nelfinavir, Saquinavir

   G. High dose Methotrexate (≥1000 mg/m2)

   H. Digoxin

   I. Cefditoren, Cefuroxime

   J. Levoketoconazole

   K. St John's Wort

   L. Bromopride, Metoclopramide

   M. Other anti-cancer therapies (chemotherapy, radiotherapy, immunotherapy, targeted therapy, hormone therapy, etc. other than the IP) which could impact the efficacy results during the study (However, local radiotherapy to alleviate ostalgia, bronchial obstruction, skin lesion, etc. are permitted. The total irradiation dose must be within the site-specific reference range for palliative therapy, and irradiation sites must be excluded from the tumor assessment.)

   N. Requiring continued treatment with systemic corticosteroids at a dose of prednisone >10 mg/day or equivalent (with exceptions of topical use such as intra-articular, intranasal, intraocular, and inhalational administration and temporary use for treatment and prevention of allergic reactions to a contrast agent or AEs [e.g., vomiting])
4. Pregnant or lactating women, or women of childbearing potential and men who are unwilling to remain abstinent or use adequate methods of contraception* during the study and for 3 months after IP administration

   * Adequate methods of contraception:
   * Hormonal contraceptives
   * Placement of an intrauterine device or intrauterine system
   * Surgical sterilization (vasectomy, tubal ligation, etc.)
5. Received/Used another investigational agent/device within 4 weeks (or 5 half-lives) prior to screening
6. Ineligibility or inability to participate in the study in the judgment of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
DLT(dose limiting toxicity) | Until 28 days from the first IP administration
  DLTs will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) ver. 5.0, and defined as CTCAE Grade ≥3 ADR(Adverse Drug Reaction)s.
AEs(Adverse Events) | Through study completion, an average of 5 months
  Any clinically significant medical condition or abnormality observed after IP administration will be collected as an AE.
Laboratory tests | Through study completion, an average of 5 months
  For collected laboratory test results, changes between before and after IP administration and/or changes in normality/abnormality will be assessed.
Vital signs | Through study completion, an average of 5 months
  For collected vital signs results, changes between before and after IP administration and/or changes in normality/abnormality will be assessed.
ECG(Electrocardiogram) | Through study completion, an average of 5 months
  ECG results will be assessed and recorded as normal or abnormal, and any clinically significant changes will be recorded as AEs in the CRF.

OTHER OUTCOMES:
AUClast | Day 1: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  AUClast of KN510 and KN713
AUCinf | Day 1: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  AUCinf of KN510 and KN713
Cmax | Day 1: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Cmax of KN510 and KN713
Tmax | Day 1: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Tmax of KN510 and KN713
CL/F | Day 1: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  CL/F of KN510 and KN713
Vd/F | Day 1: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Vd/F of KN510 and KN713
t1/2 | Day 1: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  t1/2 of KN510 and KN713
AUCtau,ss | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  AUCtau,ss of KN510 and KN713
Cmax,ss | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Cmax,ss of KN510 and KN713
Cmin,ss | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Cmin,ss of KN510 and KN713
Cav,ss | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Cav,ss of KN510 and KN713
peak-trough fluctuation (PTF) | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  peak-trough fluctuation (PTF) of KN510 and KN713
Tmax,ss | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Tmax,ss of KN510 and KN713
CLss/F | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  CLss/F of KN510 and KN713
Vd,ss/F | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  Vd,ss/F of KN510 and KN713
t1/2,ss | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  t1/2,ss of KN510 and KN713
accumulation ratio | Day 22: 0(pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post-dose
  accumulation ratio of KN510 and KN713
Objective response rate (ORR)* | Through study completion, an average of 5 months
  Proportion of subjects with best overall response (BOR) of complete response (CR) or partial response (PR) *ORR = CR + PR
Disease control rate (DCR)** | Through study completion, an average of 5 months
  Proportion of subjects with BOR of CR, PR or stable disease (SD)
  **DCR = CR + PR + SD
Exploratory Efficacy Endpoints [DOR] | 6 and 12 months
  Time from initial assessment of confirmed CR or PR to initial assessment of confirmed PD
Progression free survival (PFS) | 6 and 12 months
  Time from the start of IP treatment to PD per RECIST v1.1 or death from any cause, whichever occurs first
Overall survival (OS) | 6 and 12 months
  Time from the start of IP treatment to death from any cause
Target tumor size | Through study completion, an average of 5 months
  Maximum percentage change in the sum of longest diameters of target lesions

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, South Korea